CLINICAL TRIAL: NCT01135225
Title: EVOLVE: A Prospective Randomized Multicenter Single-blind Non-inferiority Trial to Assess the Safety and Performance of the Evolution Everolimus-Eluting Monorail Coronary Stent System (Evolution Stent System) for the Treatment of a De Novo Atherosclerotic Lesion
Brief Title: Non-inferiority Trial to Assess the Safety and Performance of the Evolution Coronary Stent
Acronym: Evolve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2060
Record Dates: First submitted 2010-05-31; First posted 2010-06-02 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stent; Percutaneous coronary intervention; Stent implantation; Evolution Stent System; Biodegradable polymer coating; Feasibility study
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PROMUS(TM) Element(TM) Coronary Stent (Active Comparator): PROMUS(TM) Element(TM) Everolimus-Eluting Coronary Stent System
  Interventions: Device: PROMUS(TM) Element (TM) Stent System
- Evolution Coronary Stent A (Experimental): Evolution Everolimus-Eluting Monorail Coronary Stent System
  Interventions: Device: Evolution Stent System
- Evolution Coronary Stent B (Experimental): Evolution Everolimus-Eluting Monorail Coronary Stent System
  Interventions: Device: Evolution Stent System

INTERVENTIONS:
Device: PROMUS(TM) Element (TM) Stent System — The PROMUS Element Everolimus-Eluting Coronary Stent System is a device/drug combination product composed of two components: a device (coronary stent system) and a drug product (a formulation of everolimus contained in a polymer coating.
  Arms: PROMUS(TM) Element(TM) Coronary Stent
Device: Evolution Stent System — The Evolution Everolimus-Eluting Monorail Coronary Stent System is a device/drug combination comprised of two regulated components: a device (coronary stent stent) and a drug product (a formulation of everolimus contained in a biodegradable polymer coating).
  Arms: Evolution Coronary Stent A; Evolution Coronary Stent B

SUMMARY:
The purpose of the EVOLVE Trial is to assess the safety and performance of the everolimus-eluting Evolution stent for the treatment of a de novo atherosclerotic lesion of up to 28 mm in length in a native coronary artery 2.25 mm to 3.5 mm in diameter. The safety and performance of two different drug release rate formulations of the Evolution Stent will be compared to the commercially available PROMUS (TM) Element (TM) drug-eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient has symptomatic coronary artery disease or documented silent ischemia
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG)
* Patient has a left ventricular ejection fraction (LVEF) ≥30% as measured within 60 days prior to enrollment
* Patient is willing to comply with all protocol-required follow-up evaluations

Exclusion Criteria:

* Patient has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute MI
* Patient with unstable angina or recent MI (within 72 hours) must have CK/CK-MB or troponin documented prior to the procedure and are excluded if any of the following criteria are met at the time of the index procedure:

  1. If CK MB >2× upper limit of normal (ULN), the patient is excluded regardless of the CK Total.
  2. If CK Total >2× ULN, either CK-MB or troponin must be drawn and the patient is excluded if either CK-MB or troponin is abnormal.
  3. If neither CK Total or CK MB is drawn but troponin is, the patient is excluded if:

     * Troponin >1× ULN and the patient has at least one of the following:
     * Patient has ischemic symptoms and ECG changes indicative of ongoing ischemia (e.g., >1 mm ST segment elevation or depression in consecutive leads or new left bundle branch block [LBBB])
     * Development of pathological Q waves in the ECG; or;
     * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality Note: Patients with stable angina must have CK/CK-MB or troponin drawn prior to the index procedure. However, the results for these patients do not need to be available prior to the index procedure and there are no exclusion criteria based on these studies.
* Patient has received an organ transplant or is on a waiting list for an organ transplant
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Patient is receiving oral or intravenous immunosuppressive therapy (e.g., inhaled steroids are not excluded ) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
* Patient is receiving chronic (≥72 hours) anticoagulation therapy (e.g., heparin, coumadin) for indications other than acute coronary syndrome
* Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Patient has a white blood cell (WBC) count <3,000 cells/mm3
* Patient has documented or suspected liver disease, including laboratory evidence of hepatitis
* Patient is on dialysis or has known renal insufficiency (e.g. serum creatinine level >2.0 mg/dL)
* Patient has active peptic ulcer disease, an active gastrointestinal (GI) bleed, other bleeding diathesis or coagulopathy, or will refuse transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Target vessel (including side branches) has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to the index procedure
* Target vessel has been treated within 10 mm proximal or distal to the target lesion (by visual estimate) with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) at any time prior to the index procedure
* Non-target vessel (including side branches) has been treated with any type of PCI (e.g., balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to the index procedure Note: 1 lesion in a non-target vessel may be treated during the index procedure prior to the treatment of the target (study) lesion. The treatment of lesion(s) in non-target vessels more than 24 hours prior to the procedure does not preclude the treatment of an additional non-target lesion during the index procedure. For example, a patient could have an RCA lesion treated 7 days prior to the index procedure and then have a non-target lesion in the LCx and a target lesion in the LAD treated during the index procedure.
* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter immediately prior to stent placement
* Planned PCI or CABG after the index procedure
* Patient previously treated at any time with coronary intravascular brachytherapy
* Patient has a known allergy to the trial stent system or protocol-required concomitant medications (e.g., stainless steel, platinum, chromium, nickel, tungsten, acrylic, fluoropolymers, everolimus, thienopyridines, aspirin, contrast) that cannot be adequately premedicated
* Patient has one of the following.

  * Other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Patient is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Patient intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Patient with known intention to procreate within 12 months after the index procedure. (Women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.)
* Patient is a woman who is pregnant or nursing. (A pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential.)
* Patient has more than 1 target lesion and 1 non-target lesion that will be treated during the index procedure

Angiographic Inclusion criteria (Visual Estimate):

* Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥ 2.25 mm and ≤3.5 mm.
* Target lesion length must be ≤ 28 mm (by visual estimate)
* Target lesion must have visually estimated stenosis ≥50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow >1.
* Target lesion must be successfully pre-dilatated.

Angiographic Exclusion criteria (visual estimate):

* Target lesion meets any of the following criteria.

  * Left main location
  * Located within 5 mm of the origin of the left anterior descending (LAD), left circumflex (LCX) or RCA by visual estimate
  * Located within a saphenous vein graft or an arterial graft
  * Will be accessed via a saphenous vein graft or arterial graft
  * Involves a side branch ≥2.0 mm in diameter by visual estimate
  * Involves a side branch <2.0 mm in diameter by visual estimate which requires treatment
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
  * Excessive tortuosity proximal to or within the lesion
  * Excessive angulation proximal to or within the lesion
  * Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
  * Restenotic from previous intervention
  * Thrombus, or possible thrombus, present in the target vessel
  * Target lesion cannot be covered by a single study stent
* Patient has unprotected left main coronary artery disease (>50% diameter stenosis)
* Patient has protected left main coronary artery disease and a target lesion in the LAD or LCX
* Patient has an additional clinically significant lesion(s) in the target vessel for which an intervention within 12 months after the index procedure may be required
* Non-target lesion to be treated during the index procedure meets any of the following criteria.

  * Located within the target vessel
  * Located within a bypass graft (venous or arterial)
  * Left main location
  * Chronic total occlusion
  * Involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
  * Requires additional unplanned stents
  * Treatment not deemed a clinical angiographic success
  * Treatment not completed prior to treatment of target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Composite safety endpoint of Target Lesion Failure (TLF) at 30 days post-procedure | 30 days
  Composite safety endpoint of Target Lesion Failure (TLF) at 30 days post-procedure:
  * Cardiac Death related to target vessel
  * Target Vessel Myocardial Infarction (TV-MI)
  * Target Lesion Revascularization (TLR)
In-stent late loss at 6 month post-procedure | 6 months post-procedure
  In-stent late loss at 6 months post-procedure measured by Quantitative Coronary Angiography (QCA)

SECONDARY OUTCOMES:
Target lesion revascularization (TLR) rate at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
Target vessel revascularization (TVR) rate at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
Target lesion failure (TLF) rate at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
Target vessel failure (TVF) rate at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
Cardiac death rate at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
Non-cardiac death rate at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
MI rate (TV and overall)at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years
Stent thrombosis rate (by Academic Research Consortium [ARC] definition)at 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years | 30 days, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, Prof, Principal Investigator — Monash Medical Centre; Stefan Verheye, Dr, Principal Investigator — AZ Middelheim
Locations (29):
- Australia (4):
  - The Prince Charles Hospital, Chermside
  - Monash Medical Centre, Clayton
  - St. Vincent's Hospital (Melbourne), Fitzroy
  - Fremantle Hospital, Fremantle
- Belgium (4):
  - Academisch Ziekenhuis Middelheim, Antwerp
  - Ziekenhuis Oost Limburg, Genk
  - UZ Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire Sart Tilman Liège, Liège
- Denmark (2):
  - Skejby Sygehus, Aarhus
  - Rigshospitalet Thoraxkirurgisk Klinik RT, Copenhagen
- France (4):
  - Polyclinique Les Fleurs, Ollioules
  - Hôpital Cochin, Paris
  - Hôpital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- New Zealand (3):
  - Dunedin Hospital, Dunedin
  - Middlemore Hospital, Otahuhu
  - North Shore Hospital, Takapuna
- Szpital Uniwersytecki im. dr. Antoniego Jurasza w Bydgoszczy, Bydgoszcz, Poland
- Spain (4):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
- Sweden (2):
  - Falu lasarett, Falun
  - Uppsala Akademiska Hospital, Uppsala
- United Kingdom (5):
  - Royal Victoria Hospital, Belfast
  - Papworth Hospital, Cambridge
  - Golden Jubilee National Hospital, Clydebank
  - Liverpool Heart and Chest Hospital, Liverpool
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Meredith IT, Verheye S, Weissman NJ, Barragan P, Scott D, Valdes Chavarri M, West NE, Kelbaek H, Whitbourn R, Walters DL, Kubica J, Thuesen L, Masotti M, Banning A, Sjogren I, Stables RH, Allocco DJ, Dawkins KD. Six-month IVUS and two-year clinical outcomes in the EVOLVE FHU trial: a randomised evaluation of a novel bioabsorbable polymer-coated, everolimus-eluting stent. EuroIntervention. 2013 Jul;9(3):308-15. doi: 10.4244/EIJV9I3A52. PMID 23872647
- [Derived] Meredith IT, Verheye S, Weissman NJ, Barragan P, Scott D, Chavarri MV, West NE, Kelbaek H, Whitbourn R, Walters DL, Kubica J, Thuesen L, Masotti M, Banning A, Sjogren I, Stables RH, Allocco DJ, Dawkins KD. Six-month IVUS and two-year clinical outcomes in the EVOLVE FHU trial: a randomised evaluation of a novel bioabsorbable polymer-coated, everolimus-eluting stent. EuroIntervention. 2013 May 22:20130416-02. Online ahead of print. PMID 23688934
- [Derived] Meredith IT, Verheye S, Dubois CL, Dens J, Fajadet J, Carrie D, Walsh S, Oldroyd KG, Varenne O, El-Jack S, Moreno R, Joshi AA, Allocco DJ, Dawkins KD. Primary endpoint results of the EVOLVE trial: a randomized evaluation of a novel bioabsorbable polymer-coated, everolimus-eluting coronary stent. J Am Coll Cardiol. 2012 Apr 10;59(15):1362-70. doi: 10.1016/j.jacc.2011.12.016. Epub 2012 Feb 15. PMID 22341736